CLINICAL TRIAL: NCT03160248
Title: An Investigator-initiated, Randomized, Double-blind, Placebo Controlled Study of Apremilast to Demonstrate Efficacy in Subjects With Nummular Eczema
Brief Title: An Investigator-initiated Study of Apremilast to Demonstrate Efficacy Nummular Eczema
Acronym: APREMINUM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP-CL-ECZ-PI-006539
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2020-10

CONDITIONS: Nummular Eczema; Eczema; Dermatitis Eczema; Nummular Dermatitis
MeSH Terms: conditions — Eczema | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Apremilast (Experimental): Patients randomized to this arm will start Apremilast with a titration phase of 5 days, followed by 30 mg Apremilast tablets twice daily (BID) by mouth (PO) for a total of 32 weeks (including titration phase).
  Interventions: Drug: Apremilast
- Placebo + Apremilast (Experimental): Patients randomized to this arm will receive identically matching placebo (including the titration phase) by mouth for first 16 weeks. Placebo participants will be switched to receive Apremilast 30 mg BID from beginning of Week 17 for another 16 weeks. In this arm Apremilast will be started without titration.
  Interventions: Drug: Apremilast; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Apremilast — This study aims on investigating the efficacy of Apremilast in nummular eczema patients.
Drug: Placebo Oral Tablet — This study aims on investigating the efficacy of Apremilast in nummular eczema patients - placebo controlled
  Arms: Placebo + Apremilast

SUMMARY:
This is an investigator-initiated, single-center, prospective, randomized, double-blind, interventional phase IIb study. Forty patients with clinically and histologically confirmed nummular eczema will be enrolled according to inclusion and exclusion criteria. Patients will be included after written informed consent is obtained. Prior to randomization, average application rate of class II topical steroids per day will be measured for 4 weeks. Subsequently, patients will be randomized in a 1:1 ratio into one arm to receive Apremilast 30 mg BID (following titration phase) for 16 weeks or a second arm receiving identically matching placebo for 16 weeks. From beginning of week 17, all patients will start an open-label treatment with Apremilast 30 mg BID until week 32. Concomitant use of topical steroids (class II) is allowed during the study. During the treatment period both placebo and Apremilast will be applied p.o. from week 0 until week 32.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically confirmed diagnosis of nummular eczema
2. Biopsy-proven, meaning histology consistent with eczema (including PAS-staining)
3. PGA ≥ 3 on a 5 point scale
4. History of continuous use of topical steroids for the last 8 weeks
5. Age 18-85 years of age, body weight ≥ 40 kg and ≤ 160 kg
6. Signed informed consent from patient

Exclusion Criteria:

1. Permanent severe diseases, especially those affecting the immune system
2. Pregnancy or breast feeding
3. History or presence of epilepsy, significant neurological disorders, depression, suicidal ideation and behaviour, cerebrovascular attacks or ischemia
4. History or presence of myocardial infarction or cardiac arrhythmia which requires drug therapy
5. Evidence of severe renal dysfunction defined as:

   * eGFR < 30 ml/min/1,73 m2 (calculated using the MDRD formula) at screening (Visit 1)
6. Evidence of significant hepatic disease defined as:

   At screening (Visit 1):
   * Alkaline phosphatase >3x upper limit of normal (ULN) or alkaline phosphatase >2,5x ULN and total bilirubin > 2xULN or
   * Aspartate transaminase (AST, SGOT]) and alanine transaminase (ALT, SGPT]) > 2.5x upper limit of normal (ULN)
7. History of lymphoproliferative disorders
8. Patients who are considered potentially unreliable or where it is envisaged the patient may not consistently attend scheduled study visits
9. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant unless they use effective contraception during the study and for 4 weeks after study completion or discontinuation. The chosen form of birth control must be effective by the time the patient receives her first dose of study drug.
10. Inability or unwillingness to undergo repeated venipuncture (e.g., because of poor tolerability or lack of access to veins)
11. Inability or unwillingness to undergo repeated punch biopsies
12. History of allergy to any component of the study medication
13. Current use of strong cytochrome P450 enzyme inducers (eg, rifampicin, phenobarbital, carbamazepine, phenytoin and St John's wort)
14. Patients with rare hereditary problems of galactose intolerance, lapp lactase deficiency or glucose-galactose malabsorption
15. Evidence of acute contact dermatitis at screening
16. Evidence of underweight, defined as BMI < 18,5 kg/m2
17. Evidence of Zink deficiency defined as Zink level < 20 µg/dL in serum

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
PGA | week 16
  Number of Patients Achieving an Improvement (Decrease) in PGA (Physician Global Assessment) by two or more points at week 16 as compared to week 0 or achieving an absolute PGA of 0 or 1 at Week 16

SECONDARY OUTCOMES:
EASI | week 16 and 32
  EASI 50 score at week 16 and 32 (Eczema Area and Severity Index)
Transepidermal Waterloss (TEWL) | week 16 and 32
  Change From Baseline in Transepidermal Waterloss (TEWL) at week 16 and 32
Histology | week 16
  Significant histological improvement at week 16 - Assessed by reduction of epidermal thickness > 30% or reduction of inflammatory infiltrate > 50 % compared to histological findings on baseline.
Use of topical steroids | week 16 and 32
  Change From Baseline in the Reduction of the Use of Topical Steroids at week 16 and 32
  - Prior to randomization and during the treatment, average application rate of class II topical steroids per day will be calculated. Participants will receive "prednicarbate" from the study centre. On each visit the tube will be weighed to measure usage.
PGA score Arm 2 | week 32
  Change in PGA score compared to baseline and week 16 for patients in Arm 2 at week 32
  - Comparison of the first and the second 16 weeks of the trial in terms of the change in PGA score from baseline for patients in Arm 2
DLQI | week 16 and 32
  Change From Baseline in the Dermatology Life Quality Index (DLQI) Total Score at Week 16 and 32
Pruritus Visual Analog Scale (VAS) | week 16 and 32
  Change From Baseline in Pruritus Visual Analog Scale (VAS) Score at Week 16 and 32
TSQM | week 16 and 32
  Change From Baseline in the Global Satisfaction Subscale of the Treatment Satisfaction Questionnaire for Medication (TSQM) Score at Week 16 and 32
Safety: Safety of Apremilast will be Assessed by Evaluating Adverse Events (AEs) - Type, frequency, severity, and relationship of the AEs to apremilast | week 36
  Safety of Apremilast will be Assessed by Evaluating Adverse Events (AEs) - Type, frequency, severity, and relationship of the AEs to apremilast

OTHER OUTCOMES:
Exploratory endpoint: Change From Baseline in metabolic functions at Week 16 and 32 - weight | week 16 and 32
  Assessed via physical examination (weight (kg))
Exploratory endpoint: Change From Baseline in metabolic functions at Week 16 and 32 - BMI | week 16 and 32
  Assessed via physical examination (BMI (kg/m2))
Exploratory endpoint: Change From Baseline in metabolic functions at Week 16 and 32 - abdominal girth | week 16 and 32
  Assessed via physical examination (abdominal girth (cm)))
Exploratory endpoint: Change From Baseline in metabolic functions at Week 16 and 32 - serum parameters | week 16 and 32
  Assessed via serum parameters (glucose, HbA1c, cholesterol, HDL, LDL, Lipoprotein (a))
Exploratory endpoint: Change From Baseline in metabolic functions at Week 16 and 32 - characterization of molecular (gene expression profil) | week 16 and 32
  Changes in metabolic functions during treatment with Apremilast vs. Placebo in the skin (biopsies at week 0 and week 16) as determined by RNA sequencing (RNAseq).

CONTACTS AND LOCATIONS:
Overall Officials: Kilian Eyerich, Principal Investigator — Technical University Munich
Locations (1):
- Technical University Munich - Department of Dermatology, Munich, Bavaria, Germany